CLINICAL TRIAL: NCT03719053
Title: Single Observed Dose Administration of Truvada® to Establish Single Dose Pharmacokinetic Standards in Healthy Individuals
Brief Title: Single Dose Truvada Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00174702
Record Dates: First submitted 2018-10-23; First posted 2018-10-25 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Medication Adherence; HIV Prevention
MeSH Terms: conditions — Medication Adherence | interventions — Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Truvada (Experimental): single oral dose of Truvada® (300 mg tenofovir disoproxil fumarate)
  Interventions: Drug: Tenofovir

INTERVENTIONS:
Drug: Tenofovir — pre- and post-dosing measurements of TFV and TFV-DP in plasma and PBMCs.
  Other Names: Truvada

SUMMARY:
This study examines tenofovir (TFV) drug concentrations in adults one day after taking a single dose of Truvada® - a pill used to prevent and treat HIV infection. The results of this study will be used to improve the (efficacy/accuracy) of a white coat adherence (WCA) detection test - a blood test that can be used to indicate medication adherence. Participants will receive one dose of Truvada®, and provide 2 total samples of blood.

DETAILED DESCRIPTION:
To establish the plasma and peripheral blood mononuclear cells (PBMC) concentrations of TFV and TFV diphosphate (TFV-DP), respectively, following a single oral dose of Truvada® [300 mg tenofovir disoproxil fumarate (TDF) in fixed dose combination with emtricitabine (FTC)], the same formulation used for HIV pre-exposure prophylaxis (PrEP), and in prior benchmarking adherence studies (HPTN 066). This will be compared to steady-state TFV and TFV-DP concentrations to more robustly differentiate single dose concentrations from steady-state concentrations.

This is part of a larger project to determine the frequency of white coat adherence in several clinical studies where doses are not observed. For purposes of diagnosing WCA with TDF, the investigators define WCA quantitatively as taking a single dose of TDF preceded by no doses in the prior week. The investigators will compare TFV and TFV-DP concentrations following an observed single oral dose of TDF/FTC to steady-state concentrations of TFV and TFV-DP after daily dosing under observation.

The study plan involves a screening visit to assess eligibility, followed by two study visits. Visit one involves pre-dose blood testing, followed by a single dose of Truvada. Visit two occurs 24-hours after visit one, and involves collection of a final post-dose blood sample. Blood will be assessed for tenofovir and tenofovir analyte concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy with no acute medical illness
* Willing to provide written informed consent
* Age 18 years of age or older
* Negative qualitative urine pregnancy test at screening and on day of dosing, prior to dosing, female participants only
* HIV-1 negative at screening, as documented by Combo Ag/Ab HIV-1/HIV-2 immunoassay
* At screening, no evidence of hepatic or renal impairment [creatinine clearance > 60 ml/min, total bilirubin ≤ upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 1.5 ULN]

Exclusion Criteria:

* Concomitant antiretroviral or other medication use, for which there is a known risk of pharmacokinetic or pharmacodynamic drug interactions.
* Active medical or psychological condition that, in the opinion of the investigator, might put the volunteer at undue risk or interfere with the participation of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Plasma Tenofovir (TFV) concentration in ng/mL | 24 hours
Peripheral Blood Mononuclear Cells (PBMC) TFV diphosphate (TFV-DP) concentration in femtomole per million cells (fmol/10^6) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hendrix, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States